CLINICAL TRIAL: NCT01999855
Title: Evaluation of the Frequency of Dysphonia by Subjective and Objective Methods in Asthmatic Patients
Brief Title: Frequency of Dysphonia in Asthmatic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: technical problem
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5517
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2017-09

CONDITIONS: Asthmatic Patients and Control Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): * the Phonatory Maximum Time
  * Vocal Handicap Index
  * Scale GRBAS of Hirano
  * Videolaryngoscopy
  Interventions: Other: Phoniatric tests
- Asthmatic patients (Experimental): * The Phonatory Maximum Time
  * Vocal Handicap Index
  * Scale GRBAS of Hirano
  * Videolaryngoscopy
  Interventions: Other: Phoniatric tests

INTERVENTIONS:
Other: Phoniatric tests
  Other Names: - the Phonatory Maximum Time; - Vocal Handicap Index; - Scale GRBAS of Hirano; - Videolaryngoscopy

SUMMARY:
For many years, it is known that asthmatics have more often dysphonia. However, no study has so far analyzed the reality of dysphonia in asthmatic by making phoniatric tests.

The etiology of dysphonia in asthmatic remains controversial. Indeed, for a long time, inhaled corticosteroids have been considered as responsible for organic abnormalities of the vocal cords. We hypothesized that women with asthma have more often dysphonia, and that dysphonia is rather functional origin.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged between 18 to 65 years
* Patient who signed the informed consent.
* affiliated with a social security system.

Patients with asthma (GINA criteria)

- persistent asthma with inhaled corticosteroids.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evidence of dysphonia. The patient will be considered as having a dysphonia if at least one of the tests (Voice Handicap Index, Rank Rough Breathy Asthenic Strained GRBAS, Quotien Phonatoire QP and Fundamental laryngeal F0) is abnormal | Four week

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric De Blay, Pr, Principal Investigator — Pôle de Pathologie Thoracique- Hôpitaux Universitaires Strasbourg
Locations (1):
- Service de pneumologie, d'allergologie et de pathologie de l'environnement, Strasbourg, France